CLINICAL TRIAL: NCT03310021
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Andexanet Alfa Administered to Healthy Japanese and Caucasian Subjects
Brief Title: A Healthy Volunteer Pharmacokinetics (PK)/Pharmacodynamics (PD), Safety and Tolerability Study of Andexanet in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-508
Record Dates: First submitted 2017-09-07; First posted 2017-10-16 (Actual); Results first posted 2020-08-14 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — PRT064445; Injections, Intravenous; apixaban; Rivaroxaban; edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind (Participant, Care Provider, Investigator, Sponsor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (Experimental): Apixaban + low dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Apixaban; Drug: Placebo
- Cohort 2 (Experimental): Rivaroxaban + high dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Rivaroxaban; Drug: Placebo
- Cohort 3 (Experimental): Edoxaban + high dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Edoxaban; Drug: Placebo
- Cohort 4 (Experimental): Edoxaban + high dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Edoxaban; Drug: Placebo
- Cohort 5 (Experimental): Apixaban + low dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Apixaban; Drug: Placebo
- Cohort 6 (Experimental): Apixaban + high dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Apixaban; Drug: Placebo
- Cohort 7 (Experimental): Edoxaban + low dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Edoxaban; Drug: Placebo
- Cohort 8 (Experimental): Apixaban + low dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Apixaban; Drug: Placebo
- Cohort 9 (Experimental): Rivaroxaban + low dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Rivaroxaban; Drug: Placebo
- Cohort 10 (Experimental): Edoxaban + low dose andexanet
  Interventions: Biological: Andexanet alfa; Drug: Edoxaban; Drug: Placebo

INTERVENTIONS:
Biological: Andexanet alfa — fXa inhibitor antidote
  Other Names: 200 mg/vial for IV injection
Drug: Apixaban — factor Xa inhibitor
  Other Names: Eliquis
  Arms: Cohort 1; Cohort 5; Cohort 6; Cohort 8
Drug: Rivaroxaban — factor Xa inhibitor
  Other Names: Xarelto
  Arms: Cohort 2; Cohort 9
Drug: Edoxaban — factor Xa inhibitor
  Other Names: Savaysa, Lixiana
  Arms: Cohort 10; Cohort 3; Cohort 4; Cohort 7
Drug: Placebo — Placebo

SUMMARY:
"This is a single-center, randomized, double-blind, and placebo-controlled trial designed to: 1) demonstrate the degree to which administered andexanet doses can reverse Factor Ten A (FXa)-inhibitor induced anticoagulation; and 2) evaluate the safety and PK/PD of andexanet in healthy Japanese subjects taking direct FXa inhibitors at therapeutic doses."

ELIGIBILITY:
Inclusion Criteria:

1. Must be in reasonably good health as determined by the Investigator based on medical history, full physical examination (including blood pressure and pulse rate measurement), 12-lead ECG, and clinical laboratory tests. Subjects with well-controlled, chronic, stable conditions (e.g., controlled hypertension, non-insulin dependent diabetes, osteoarthritis, hypothyroidism) may be enrolled based on the clinical judgment of the Investigator.
2. For all cohorts except Cohort 5, subjects must be of Japanese ethnicity, defined as having four ethnic Japanese grandparents. Subjects may not have lived outside of Japan for more than 10 years. For Cohort 5, subjects must be of Caucasian race.
3. Must be between the ages of 18 and 75 years, inclusive, at the time of signing of the Inform Consent Form (ICF).
4. Agrees to have any dietary or nutritional supplements reviewed by the Investigator and potentially held during the study if advised by the Investigator. Standard multivitamin and mineral supplementation will be permitted.
5. Agrees to comply with the contraception and reproduction restrictions of the study:

   * Men whose sexual partner is of childbearing potential and/or who are not monogamous must be using two acceptable methods of contraception, at least one of which must be a barrier method (e.g., spermicidal gel plus condom), for the entire duration of the study and for at least 1 month following study-drug administration; and men must refrain from attempting to father a child or donating sperm in the 1 month following the study-drug administration. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
   * Men who report surgical sterilization (e.g., bilateral vasectomy) must have had the procedure at least 6 months before study drug administration.
   * Surgical sterilization procedures should be supported with clinical documentation and noted in the Relevant Medical History/Current Medical Conditions section of the case report forms (CRFs).
   * Women of childbearing potential must be using two medically acceptable methods of contraception, at least one of which must be a barrier method (e.g., non-hormone containing intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom), from the time of Screening and for the duration of the study, through at least 1 month following study drug administration. Note: Oral and topical hormonal contraceptive use, as well as the use of hormone-containing intra-uterine devices, is not permitted due to their increased risk of thromboembolism. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post- ovulation methods) and withdrawal are not acceptable methods of contraception; OR
   * Postmenopausal women must have had no regular menstrual bleeding for at least 1 year before initial dosing and either be over the age of 60 years or have an elevated plasma follicle-stimulating hormone (FSH) level (i.e., > 40 milli-international units (mIU)/mL) at Screening;
   * Women who report surgical sterilization (i.e., hysterectomy, tubal ligation, and/or bilateral oophorectomy) must have had the procedure at least 6 months before study drug administration. Surgical sterilization procedures should be supported with clinical documentation and noted in the Relevant Medical History/Current Medical Conditions section of the CRF; AND All female subjects must have a documented negative pregnancy test result at Screening and on Study Day -1.
6. Systolic blood pressure < 160 mmHg and diastolic blood pressure < 90 mmHg at Screening and Day -1.
7. The following laboratory values must be within the normal laboratory reference range within 45 days of Day -1: Prothrombin Time (PT), Activated Partial Thromboplastin Time (aPTT), and Activated Clotting Time (ACT); hemoglobin, hematocrit, and platelet count.
8. The following laboratory values must be equal to or below 2 times the upper limit of normal (ULN) range within 45 days of Day -1: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and total bilirubin.
9. The Screening serum creatinine must be below 1.5 mg/dL within 45 days of Day -1.
10. Body mass index of less than 30 kg/m2, inclusive, and body weight between 50 kg and 80 kg, inclusive. In addition, subjects must be greater than 60 kg for Cohorts 3, 4, and 10.
11. Agrees to abstain from alcohol consumption for the duration of the domicile period, and from the use of drugs of abuse for the duration of the study.
12. Able to read and give written informed consent and has signed a consent form approved by the Investigator's Institutional Review Board (IRB) or Independent Ethics Committee (IEC)."

Exclusion Criteria:

1. Previous use of andexanet or previous participation in the current study (even if the subject received placebo).
2. History of abnormal bleeding, signs or symptoms of active bleeding, or risk factors for bleeding.
3. Has a stool specimen that was positive for occult blood within 6 months of study Screening or during the Screening Period.
4. Past or current medical history of thrombosis, any sign or symptom that suggests an increased risk of a systemic thrombotic condition or thrombotic event, or recent events that may increase risk of thrombosis.

   a. For example, subjects with a known or suspected hypercoagulable state, history of Venous Thromboembolism(VTE), Deep Venous Thrombosis (DVT), stroke, myocardial infarction (MI), cancer (other than non-melanoma skin cancer), atrial fibrillation, heart failure, cardiomyopathy, phlebitis, lower extremity edema, major surgery, or trauma within 2 months of Study Day -1, airplane travel with a planned flight time for any single flight segment ≥ 6 hours during the 4 weeks prior to Study Day -1, or general immobility are excluded.
5. Absolute or relative contraindication to anticoagulation or treatment with apixaban, rivaroxaban, and/or edoxaban.
6. Prior consumption of (by any route) one or more doses of aspirin (including baby aspirin), salicylate or subsalicylate, other antiplatelet drugs (e.g., ticlopidine, clopidogrel), non-steroidal anti-inflammatory drugs, fibrinolytic, or any anticoagulant within 7 days prior to Day -1 or is anticipated to require such drugs during the study.
7. Receipt of (by any route) hormonal contraception, post- menopausal hormone replacement therapy (HRT) (including over-the-counter products), or testosterone during the 4 weeks prior to Study Day -1 or is anticipated to require such drugs during the study.
8. Family history of or risk factors for a hypercoagulable or thrombotic condition, including one of the following:

   1. Factor V Leiden carrier or homozygote.
   2. Protein C, S, or ATIII activity below the normal range.
9. History of adult asthma or chronic obstructive pulmonary disease or current regular or as needed use of inhaled medications.
10. Active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or HIV-1/2 infection.
11. Use of any drugs that are strong dual inhibitors or inducers of CYP3A4 (apixaban and rivaroxaban cohorts only) and P-gp (all cohorts) within 7 days prior to Study Day -1 or anticipated need for such drugs during the study.
12. Participation in an investigational drug study within 45 days of Day -1 or Day -1 is within 5 half-lives of the investigational compound.
13. Positive screen for drugs of abuse at Day -1 that is not explained by a prescription medication that the subject is known to be taking.
14. A medical or surgical condition that may impair drug (anticoagulant or andexanet) metabolism.
15. Allergy to any of the vehicle ingredients: Tris, arginine, sucrose, hydrochloric acid, mannitol, and polysorbate 80.
16. Allergy to soy or soy products.
17. Current breastfeeding or a positive pregnancy test at Screening or Day -1.
18. Any condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or interpretation of the study results, or that would in the opinion of the Investigator increase the risk of the subject's participation in the study. This would include but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy, or any unexplained blackouts.
19. The subject is not judged by the study staff to have adequate bilateral venous access.
20. Unwillingness to adhere to the activity requirements of the study."

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Subjects
Pre-assignment Details: One subject in cohort 10 (Edoxaban/Placebo) discontinued due to protocol deviation (mis-enrolled, inclusion criteria #10 not met(weight>80kg). This subject (100003) is not summarized in tables because he/she did not receive any andexanet/Placebo. The safety population (N=107) is defined as having received study drug andexanet/placebo.
Groups:
- Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet: Andexanet 400 mg bolus+4 mg/min 120 minute Andexanet infusion (dosing at 3 hours post-apixaban); Japanese Subjects
- Cohort 1 Apixaban 5 mg BID/Placebo: Placebo 400 mg bolus+4 mg/min 120 minute infusion (placebo dosing at 3 hours post-apixaban); Japanese Subjects
- Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet: Andexanet 800 mg bolus+ 8 mg/min 120 minute infusion (dosing at 4 hours post-rivaroxaban); Japanese Subjects
- Cohort 2 Rivaroxaban 15 mg BID/Placebo: Placebo 800 mg bolus+ 8 mg/min 120 minute infusion placebo (dosing at 4 hours post-rivaroxaban); Japanese Subjects
- Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet: Andexanet 800 mg bolus+8 mg/min 120 minutes infusion (dosing at 3 hours post-edoxaban); Japanese Subjects
- Cohort 3 Edooxaban 60 mg QD/Placebo: Placebo 800 mg bolus+8 mg/min 120 minutes infusion (dosing at 3 hours post-edoxaban); Japanese Subjects
- Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet: Andexanet 800 mg bolus+8 mg/min 120 minutes infusion (dosing at 90 minutes post-edoxaban); Japanese Subjects
- Cohort 4 Edooxaban 60 mg QD/Placebo: Placebo 800 mg bolus+8 mg/min 120 minutes infusion (dosing at 90 minutes post-edoxaban); Japanese Subjects
- Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet: 400 mg bolus+4 mg/min 120 minute Andexanet infusion (dosing at 3 hours post-apixaban); Caucasian Subjects
- Cohort 5 Apixaban 5 mg BID/Placebo: Placebo 400 mg bolus+4 mg/min 120 minute infusion (placebo dosing at 3 hours post-apixaban); Caucasian Subjects
- Cohort 6 Apixaban 10 mg BID/High Dose Andexanet: Andexanet 800 mg bolus+8 mg/min 120 minute infusion (dosing at 3 hours post-apixaban); Japanese Subjects
- Cohort 6 Apixaban 10 mg BID/Placebo: Placebo 800 mg bolus+8 mg/min 120 minute infusion (dosing at 3 hours post-apixaban); Japanese Subjects
- Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet: Andexanet 400 mg bolus+4 mg/min 120 minute infusion (dosing at 90 minutes post-edoxaban); Japanese Subjects
- Cohort 7 Edoxaban 30 mg QD/Placebo: Placebo 400 mg bolus+4 mg/min 120 minute infusion (dosing at 90 minutes post-edoxaban); Japanese Subjects
- Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet: Andexanet 400 mg bolus+4 mg/min 120 minute infusion (dosing at 8 hours post-apixaban); Japanese Subjects
- Cohort 8 Apixaban 10 mg BID/Placebo: Placebo 400 mg bolus+4 mg/min 120 minute infusion (dosing at 8 hours post-apixaban); Japanese Subjects
- Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet: Andexanet 400 mg bolus+4 mg/min 120 minute infusion (dosing at 8 hours post-rivaroxaban); Japanese Subjects
- Cohort 9 Rivaroxaban 15 mg BID/Placebo: Placebo 400 mg bolus+4 mg/min 120 minute infusion (dosing at 8 hours post-rivaroxaban); Japanese Subjects
- Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet: Andexanet 400 mg bolus+4 mg/min 120 minute infusion (dosing at 8 hours post-edoxaban); Japanese Subjects
- Cohort 10 Edoxaban 60 mg QD/Placebo: Placebo 400 mg bolus+4 mg/min 120 minute infusion (dosing at 8 hours post-edoxaban); Japanese Subjects
Period: Overall Study
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Started | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
Completed | 6 | 3 | 6 | 3 | 8 | 4 | 7 | 4 | 6 | 3 | 5 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis population will include all enrolled subjects who received any amount of study drug (andexanet or placebo) treatment.
  All subjects in the safety population will be associated with the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo | Total
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.00 (8.99) | 52.00 (6.56) | 46.83 (17.50) | 55.33 (12.22) | 42.38 (10.45) | 36.75 (9.32) | 33.13 (9.26) | 33.00 (7.30) | 35.00 (14.53) | 30.33 (2.08) | 44.17 (11.02) | 42.33 (12.74) | 38.13 (11.04) | 47.75 (8.96) | 42.17 (7.70) | 46.33 (12.42) | 49.70 (12.88) | 33.60 (5.13) | 30.13 (9.91) | 39.00 (6.24) | 40.69 (11.97)
Age, Continuous [Median (Full Range); unit: years] | 44.50 [32.0 to 55.0] | 51.00 [46.0 to 59.0] | 47.50 [24.0 to 67.0] | 58.00 [42.0 to 66.0] | 45.00 [29.0 to 56.0] | 35.50 [27.0 to 49.0] | 33.0 [21.0 to 50.0] | 31.50 [25.0 to 41.0] | 31.50 [21.0 to 60.0] | 31.00 [28.0 to 32.0] | 46.50 [26.0 to 55.0] | 36.00 [34.0 to 57.0] | 34.50 [23.0 to 59.0] | 47.00 [38.0 to 59.0] | 41.00 [33.0 to 53.0] | 53.00 [32.0 to 54.0] | 51.00 [28.0 to 69.0] | 35.00 [26.0 to 40.0] | 28.50 [20.0 to 48.0] | 41.00 [32.0 to 44.0] | 38.00 [20.0 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 1 | 4 | 2 | 3 | 1 | 4 | 1 | 2 | 1 | 36
  Male | 3 | 1 | 2 | 2 | 8 | 4 | 7 | 4 | 3 | 2 | 4 | 2 | 4 | 2 | 3 | 2 | 6 | 4 | 6 | 2 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
  Asian | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 0 | 0 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Anti-Fxa Activity From Baseline to the End of Infusion (EOI) Nadir.
Description: The primary efficacy endpoint is the percent change in the anti-FXa activity from baseline to the end of infusion (EOI) nadir.
Time Frame: Baseline to the end of infusion (EOI) nadir, approximately 2.5 hours
Population: Efficacy Population: all randomized subjects who received andexanet or placebo during the double-blind treatment period and had at least one evaluable post-baseline efficacy assessment as well as the required baseline sample assessment.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
percent change | -94.50 [-96.00 to -90.00] | -29.00 [-32.00 to -18.00] | -98.00 [-99.00 to -97.00] | -37.00 [-53.00 to -34.00] | -81.00 [-89.00 to -51.00] | -47.50 [-62.00 to -34.00] | -75.50 [-82.00 to -45.00] | -37.00 [-46.00 to -16.00] | -93.00 [-94.00 to -91.00] | -34.00 [-53.00 to -24.00] | -97.00 [-98.00 to -96.00] | -31.00 [-35.00 to -30.00] | -52.50 [-69.00 to -34.00] | -37.00 [-67.00 to -17.00] | -92.00 [-95.00 to -90.00] | -24.00 [-31.00 to -21.00] | -93.50 [-98.00 to -89.00] | -37.00 [-56.00 to -29.00] | -63.50 [-80.00 to -57.00] | -27.00 [-34.00 to -25.00]
Statistical Analysis 1: Comparison: Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 1 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0275, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -65.5, 95% CI 2-sided [-78.00 to -58.00]
Statistical Analysis 2: Comparison: Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet vs Cohort 2 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.025, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -61, 95% CI 2-sided [-65.00 to -44.00]
Statistical Analysis 3: Comparison: Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 3 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0136, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -32.5, 95% CI 2-sided [-47.00 to -9.00]
Statistical Analysis 4: Comparison: Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 4 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0136, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -36.5, 95% CI 2-sided [-62.00 to -9.00]
Statistical Analysis 5: Comparison: Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 5 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.025, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -59, 95% CI 2-sided [-70.00 to -38.00]
Statistical Analysis 6: Comparison: Cohort 6 Apixaban 10 mg BID/High Dose Andexanet vs Cohort 6 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0119, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -66, 95% CI 2-sided [-68.00 to -61.00]
Statistical Analysis 7: Comparison: Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet vs Cohort 7 Edoxaban 30 mg QD/Placebo; Test type: Superiority; p = 0.2667, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -15.5, 95% CI 2-sided [-38.00 to 17.00]
Statistical Analysis 8: Comparison: Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet vs Cohort 8 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0238, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -68, 95% CI 2-sided [-74.00 to -59.00]
Statistical Analysis 9: Comparison: Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet vs Cohort 9 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0007, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -56.5, 95% CI 2-sided [-65.00 to -39.00]
Statistical Analysis 10: Comparison: Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet vs Cohort 10 Edoxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0121, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -35, 95% CI 2-sided [-53.00 to -24.00]

2. Secondary Outcome: Percent Change in Anti-Fxa Activity From Baseline to the End of Bolus (EOB) Nadir.
Description: The percent change from baseline in anti-FXa activity at its end of bolus (EOB) nadir.
Time Frame: Baseline to the end of bolus (EOB) nadir, approximately 2.5 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
percent change | -94.50 [-95.00 to -92.00] | -14.00 [-15.00 to -12.00] | -97.50 [-98.00 to -96.00] | -18.00 [-29.00 to -1.00] | -65.50 [-87.00 to -8.00] | -16.00 [-46.00 to -13.00] | -22.50 [-78.00 to 0.00] | -15.00 [-19.00 to 7.00] | -94.00 [-94.00 to -92.00] | -10.00 [-21.00 to -7.00] | -96.00 [-97.00 to -95.00] | -18.00 [-21.00 to -14.00] | -58.00 [-78.00 to -1.00] | -8.00 [-13.00 to -1.00] | -94.50 [-96.00 to -93.00] | -5.00 [-16.00 to -3.00] | -95.00 [-98.00 to -93.00] | -11.00 [-28.00 to -9.00] | -73.00 [-80.00 to -61.00] | -4.00 [-12.00 to -4.00]
Statistical Analysis 1: Comparison: Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 1 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0256, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -80, 95% CI 2-sided [-83.00 to -77.00]
Statistical Analysis 2: Comparison: Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet vs Cohort 2 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.025, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -79.5, 95% CI 2-sided [-97.00 to -67.00]
Statistical Analysis 3: Comparison: Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 3 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.074, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -37, 95% CI 2-sided [-66.00 to 5.00]
Statistical Analysis 4: Comparison: Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 4 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.1066, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -10.5, 95% CI 2-sided [-59.00 to 10.00]
Statistical Analysis 5: Comparison: Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 5 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0219, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -84, 95% CI 2-sided [-87.00 to -71.00]
Statistical Analysis 6: Comparison: Cohort 6 Apixaban 10 mg BID/High Dose Andexanet vs Cohort 6 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0262, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -78, 95% CI 2-sided [-83.00 to -74.0]
Statistical Analysis 7: Comparison: Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet vs Cohort 7 Edoxaban 30 mg QD/Placebo; Test type: Superiority; p = 0.0412, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -50, 95% CI 2-sided [-65.00 to 0.00]
Statistical Analysis 8: Comparison: Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet vs Cohort 8 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0269, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -89.5, 95% CI 2-sided [-93.00 to -77.00]
Statistical Analysis 9: Comparison: Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet vs Cohort 9 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0026, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -84, 95% CI 2-sided [-86.00 to -69.00]
Statistical Analysis 10: Comparison: Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet vs Cohort 10 Edoxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0181, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -65, 95% CI 2-sided [-76.00 to -57.00]

3. Secondary Outcome: Percent Change in Free Fxa Inhibitor Concentration From Baseline to the End of Bolus (EOB) Nadir.
Description: The percent change from baseline in free FXa inhibitors concentration (ng/mL) at its EOB nadir.
Time Frame: Baseline to the end of bolus (EOB) nadir, approximately 2.5 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 9 | 5 | 8 | 3
percent change | -93.00 [-94.70 to -90.38] | -11.94 [-18.42 to -1.71] | -97.72 [-97.97 to -95.70] | -28.57 [-47.06 to -1.06] | -78.20 [-86.17 to -59.17] | -17.60 [-27.95 to -10.15] | -56.05 [-77.92 to -40.69] | -2.49 [-28.57 to 12.48] | -94.45 [-96.56 to -93.04] | 5.80 [-8.56 to 36.52] | -93.57 [-97.30 to -90.08] | -12.94 [-24.34 to -10.94] | -70.88 [-87.12 to -44.80] | -5.48 [-12.67 to 18.07] | -91.61 [-95.51 to -89.76] | -0.32 [-28.93 to 33.37] | -95.51 [-97.09 to -93.43] | -14.02 [-30.10 to -4.10] | -75.80 [-85.51 to -70.44] | -17.91 [-26.80 to 26.42]
Statistical Analysis 1: Comparison: Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 1 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -81.06, 95% CI 2-sided [-92.99 to -71.96]
Statistical Analysis 2: Comparison: Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet vs Cohort 2 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -69.15, 95% CI 2-sided [-96.91 to -48.64]
Statistical Analysis 3: Comparison: Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 3 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -57.39, 95% CI 2-sided [-72.07 to -40.03]
Statistical Analysis 4: Comparison: Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 4 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -54.96, 95% CI 2-sided [-80.42 to -25.50]
Statistical Analysis 5: Comparison: Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 5 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -100.25, 95% CI 2-sided [-133.08 to -84.48]
Statistical Analysis 6: Comparison: Cohort 6 Apixaban 10 mg BID/High Dose Andexanet vs Cohort 6 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -79.87, 95% CI 2-sided [-86.36 to -65.74]
Statistical Analysis 7: Comparison: Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet vs Cohort 7 Edoxaban 30 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -65.02, 95% CI 2-sided [-89.54 to -39.17]
Statistical Analysis 8: Comparison: Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet vs Cohort 8 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -91.29, 95% CI 2-sided [-128.88 to -60.83]
Statistical Analysis 9: Comparison: Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet vs Cohort 9 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0034, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -81.49, 95% CI 2-sided [-91.05 to -65.96]
Statistical Analysis 10: Comparison: Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet vs Cohort 10 Edoxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0189, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -58.47, 95% CI 2-sided [-110.86 to -46.12]

4. Secondary Outcome: Percent Change in Free Fxa Inhibitor Concentration From Baseline to the End of Infusion (EOI) Nadir.
Description: The percent change from baseline in free FXa inhibitors concentration (ng/mL) at its EOI nadir.
Time Frame: Baseline to the end of infusion (EOI) nadir, approximately 2.5 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
percent change | -92.940 [-94.610 to -90.400] | -33.550 [-37.780 to -28.130] | -98.650 [-99.060 to -97.610] | -39.390 [-70.670 to -28.720] | -85.005 [-93.140 to -68.740] | -48.710 [-49.790 to -38.980] | -81.040 [-89.300 to -67.660] | -42.755 [-53.330 to -25.890] | -93.495 [-96.180 to -91.240] | -31.830 [-47.460 to -20.360] | -96.65 [-97.62 to -94.80] | -29.02 [-32.81 to -20.22] | -62.72 [-76.52 to -55.03] | -24.34 [-46.86 to -11.07] | -90.63 [-91.57 to -86.02] | -31.45 [-37.88 to 9.45] | -94.89 [-97.44 to -85.09] | -37.82 [-54.92 to -36.30] | -67.10 [-81.33 to -49.62] | -34.25 [-36.17 to -15.47]
Statistical Analysis 1: Comparison: Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 1 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -59.39, 95% CI 2-sided [-66.48 to -52.62]
Statistical Analysis 2: Comparison: Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet vs Cohort 2 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -59.26, 95% CI 2-sided [-70.34 to -26.94]
Statistical Analysis 3: Comparison: Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 3 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -36.76, 95% CI 2-sided [-46.14 to -29.76]
Statistical Analysis 4: Comparison: Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 4 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -36.82, 95% CI 2-sided [-55.81 to -20.46]
Statistical Analysis 5: Comparison: Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 5 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -61.67, 95% CI 2-sided [-75.82 to -43.78]
Statistical Analysis 6: Comparison: Cohort 6 Apixaban 10 mg BID/High Dose Andexanet vs Cohort 6 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -67.63, 95% CI 2-sided [-77.40 to -61.99]
Statistical Analysis 7: Comparison: Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet vs Cohort 7 Edoxaban 30 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -40.33, 95% CI 2-sided [-59.77 to -11.17]
Statistical Analysis 8: Comparison: Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet vs Cohort 8 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -59.18, 95% CI 2-sided [-101.02 to -48.14]
Statistical Analysis 9: Comparison: Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet vs Cohort 9 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0027, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -54.63, 95% CI 2-sided [-59.14 to -41.19]
Statistical Analysis 10: Comparison: Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet vs Cohort 10 Edoxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0189, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = -38.14, 95% CI 2-sided [-65.78 to -15.37]

5. Secondary Outcome: Change in Thrombin Generation From Baseline to the End of Bolus (EOB) Nadir.
Description: The change in thrombin generation from baseline to its EOB peak.
Time Frame: Baseline to the end of bolus (EOB) nadir, approximately 2.5 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: nM.min
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
nM.min | 1145.03 [708.92 to 1538.44] | 179.94 [161.09 to 234.44] | 1337.28 [1155.95 to 1632.28] | 209.99 [57.26 to 386.49] | 758.92 [560.66 to 1494.51] | 215.71 [-15.75 to 319.23] | 815.07 [603.90 to 949.73] | 48.59 [22.87 to 165.84] | 1244.30 [1106.36 to 1714.52] | 103.13 [-22.26 to 142.33] | 1177.47 [1081.47 to 1564.10] | 0.16 [-106.20 to 92.65] | 781.42 [381.40 to 918.54] | 67.97 [-319.74 to 157.51] | 1184.62 [1038.43 to 1394.74] | 2.69 [-76.71 to 36.71] | 1306.23 [846.48 to 1442.27] | 117.50 [44.14 to 163.39] | 902.17 [582.77 to 1405.55] | -92.82 [-245.48 to 198.13]
Statistical Analysis 1: Comparison: Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 1 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 965.09, 95% CI 2-sided [474.48 to 1377.35]
Statistical Analysis 2: Comparison: Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet vs Cohort 2 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1127.29, 95% CI 2-sided [769.46 to 1575.02]
Statistical Analysis 3: Comparison: Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 3 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 574.89, 95% CI 2-sided [307.65 to 1175.28]
Statistical Analysis 4: Comparison: Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 4 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 715.34, 95% CI 2-sided [535.38 to 836.40]
Statistical Analysis 5: Comparison: Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 5 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1141.17, 95% CI 2-sided [964.03 to 1736.78]
Statistical Analysis 6: Comparison: Cohort 6 Apixaban 10 mg BID/High Dose Andexanet vs Cohort 6 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1198.83, 95% CI 2-sided [988.82 to 1670.30]
Statistical Analysis 7: Comparison: Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet vs Cohort 7 Edoxaban 30 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 721.21, 95% CI 2-sided [585.92 to 1108.92]
Statistical Analysis 8: Comparison: Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet vs Cohort 8 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1204.62, 95% CI 2-sided [1001.72 to 1471.45]
Statistical Analysis 9: Comparison: Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet vs Cohort 9 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0027, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1180.5, 95% CI 2-sided [857.21 to 1296.02]
Statistical Analysis 10: Comparison: Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet vs Cohort 10 Edoxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0189, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 976.59, 95% CI 2-sided [585.99 to 1498.37]

6. Secondary Outcome: Change in Thrombin Generation From Baseline to the End of Infusion (EOI) Nadir.
Description: The change in thrombin generation from baseline to its EOI peak.
Time Frame: Baseline to the end of infusion (EOI) nadir, approximately 2.5 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: nM.min
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 8 | 4 | 8 | 4 | 6 | 3 | 6 | 3 | 8 | 4 | 6 | 3 | 10 | 5 | 8 | 3
nM.min | 1000.630 [695.120 to 1519.850] | 171.220 [157.740 to 189.720] | 1329.580 [1161.360 to 1679.680] | 207.590 [126.910 to 287.490] | 804.405 [692.880 to 1560.300] | 347.535 [107.360 to 482.840] | 910.935 [775.950 to 1108.160] | 236.610 [126.010 to 295.710] | 1130.575 [1022.120 to 1460.710] | 118.130 [108.660 to 163.040] | 1119.41 [969.95 to 1567.02] | 108.67 [-67.28 to 150.99] | 833.46 [571.27 to 939.46] | 175.72 [-290.06 to 336.63] | 1058.09 [809.14 to 1335.39] | 138.14 [119.11 to 145.40] | 1173.38 [773.75 to 1399.21] | 293.15 [142.08 to 324.41] | 793.44 [564.56 to 1339.52] | -72.69 [-302.36 to 52.67]
Statistical Analysis 1: Comparison: Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 1 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 826.9, 95% CI 2-sided [505.40 to 1362.11]
Statistical Analysis 2: Comparison: Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet vs Cohort 2 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1125.7, 95% CI 2-sided [873.87 to 1552.77]
Statistical Analysis 3: Comparison: Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 3 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 538.84, 95% CI 2-sided [291.20 to 1077.46]
Statistical Analysis 4: Comparison: Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet vs Cohort 4 Edooxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 687.57, 95% CI 2-sided [500.92 to 902.73]
Statistical Analysis 5: Comparison: Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet vs Cohort 5 Apixaban 5 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1012.45, 95% CI 2-sided [859.08 to 1352.05]
Statistical Analysis 6: Comparison: Cohort 6 Apixaban 10 mg BID/High Dose Andexanet vs Cohort 6 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 1057.27, 95% CI 2-sided [818.96 to 1634.30]
Statistical Analysis 7: Comparison: Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet vs Cohort 7 Edoxaban 30 mg QD/Placebo; Test type: Superiority; p = 0.0085, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 630.81, 95% CI 2-sided [421.78 to 1124.28]
Statistical Analysis 8: Comparison: Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet vs Cohort 8 Apixaban 10 mg BID/Placebo; Test type: Superiority; p = 0.0282, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 925.84, 95% CI 2-sided [663.74 to 1216.28]
Statistical Analysis 9: Comparison: Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet vs Cohort 9 Rivaroxaban 15 mg BID/Placebo; Test type: Superiority; p = 0.0027, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 871.11, 95% CI 2-sided [631.67 to 1051.06]
Statistical Analysis 10: Comparison: Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet vs Cohort 10 Edoxaban 60 mg QD/Placebo; Test type: Superiority; p = 0.0189, 2-sided Wilcoxon Rank Sum; Hodges lehman Location shift = 874.44, 95% CI 2-sided [637.25 to 1412.21]

ADVERSE EVENTS:
Time Frame: Study day 1 to 39
Description: Treatment emergent AEs occurring between informed consent and the Termination Visit will be recorded on the e-CRFs. All AEs should be monitored until they are resolved, reach a level of stability and are not expected to improve further, or are clearly determined to be due to a subject's stable or chronic condition or intercurrent illness. Any AE that begins after completion of the study and that the Investigator considers to be related to study medication, must be reported to Portola.
Arm/Group | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 1 Apixaban 5 mg BID/Placebo | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet | Cohort 2 Rivaroxaban 15 mg BID/Placebo | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 3 Edooxaban 60 mg QD/Placebo | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet | Cohort 4 Edooxaban 60 mg QD/Placebo | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet | Cohort 5 Apixaban 5 mg BID/Placebo | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet | Cohort 6 Apixaban 10 mg BID/Placebo | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet | Cohort 7 Edoxaban 30 mg QD/Placebo | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet | Cohort 8 Apixaban 10 mg BID/Placebo | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet | Cohort 9 Rivaroxaban 15 mg BID/Placebo | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet | Cohort 10 Edoxaban 60 mg QD/Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 0/3 | 0/8 | 0/4 | 0/8 | 0/4 | 0/6 | 0/3 | 0/6 | 0/3 | 0/8 | 0/4 | 0/6 | 0/3 | 0/10 | 0/5 | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 0/3 | 0/8 | 0/4 | 0/8 | 0/4 | 1/6 | 0/3 | 0/6 | 0/3 | 0/8 | 0/4 | 0/6 | 0/3 | 0/10 | 0/5 | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 2/3 | 3/6 | 1/3 | 1/8 | 1/4 | 3/8 | 1/4 | 4/6 | 0/3 | 2/6 | 1/3 | 2/8 | 0/4 | 3/6 | 0/3 | 2/10 | 0/5 | 1/8 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet (N=6) | Cohort 1 Apixaban 5 mg BID/Placebo (N=3) | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet (N=6) | Cohort 2 Rivaroxaban 15 mg BID/Placebo (N=3) | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet (N=8) | Cohort 3 Edooxaban 60 mg QD/Placebo (N=4) | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet (N=8) | Cohort 4 Edooxaban 60 mg QD/Placebo (N=4) | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet (N=6) | Cohort 5 Apixaban 5 mg BID/Placebo (N=3) | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet (N=6) | Cohort 6 Apixaban 10 mg BID/Placebo (N=3) | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet (N=8) | Cohort 7 Edoxaban 30 mg QD/Placebo (N=4) | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet (N=6) | Cohort 8 Apixaban 10 mg BID/Placebo (N=3) | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet (N=10) | Cohort 9 Rivaroxaban 15 mg BID/Placebo (N=5) | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet (N=8) | Cohort 10 Edoxaban 60 mg QD/Placebo (N=3)
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | NA | NA | NA | NA | NA | NA | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Apixaban 5 mg BID/Low Dose Andexanet (N=6) | Cohort 1 Apixaban 5 mg BID/Placebo (N=3) | Cohort 2 Rivaroxaban15 mg BID/High Dose Andexanet (N=6) | Cohort 2 Rivaroxaban 15 mg BID/Placebo (N=3) | Cohort 3 Edoxaban 60 mg QD/High Dose Andexanet (N=8) | Cohort 3 Edooxaban 60 mg QD/Placebo (N=4) | Cohort 4 Edoxaban 60 mg QD/High Dose Andexanet (N=8) | Cohort 4 Edooxaban 60 mg QD/Placebo (N=4) | Cohort 5 Apixaban 5 mg BID/Low Dose Andexanet (N=6) | Cohort 5 Apixaban 5 mg BID/Placebo (N=3) | Cohort 6 Apixaban 10 mg BID/High Dose Andexanet (N=6) | Cohort 6 Apixaban 10 mg BID/Placebo (N=3) | Cohort 7 Edoxaban 30 mg QD/Low Dose Andexanet (N=8) | Cohort 7 Edoxaban 30 mg QD/Placebo (N=4) | Cohort 8 Apixaban 10 mg BID/Low Dose Andexanet (N=6) | Cohort 8 Apixaban 10 mg BID/Placebo (N=3) | Cohort 9 Rivaroxaban 15 mg BID/Low Dose Andexanet (N=10) | Cohort 9 Rivaroxaban 15 mg BID/Placebo (N=5) | Cohort 10 Edoxaban 60 mg QD /Low Dose Andexanet (N=8) | Cohort 10 Edoxaban 60 mg QD/Placebo (N=3)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter Site Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel Puncture Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03310021/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Part 1 (2018-07-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT03310021/SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Part 2 (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03310021/SAP_002.pdf